CLINICAL TRIAL: NCT04630990
Title: Effectiveness and Safety of Elagolix Treatment in Moderate to Severe Endometriosis-associated Pain in Routine Clinical Practice in Israel- ENDORSE Study
Brief Title: Study Of Oral Elagolix Tablets To Assess the Tolerability and Change in Disease Symptoms in Adult Female Participants With Moderate to Severe Endometriosis-associated Pain
Acronym: ENDORSE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-399
Record Dates: First submitted 2020-10-29; First posted 2020-11-16 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Endometriosis
Keywords: Elagolix; Orilissa; ABT-620; Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Treated With Elagolix: Participants will receive Elagolix according to the local label.

SUMMARY:
Endometriosis is an abnormal, estrogen-dependent growth of endometrial tissue outside the uterus that frequently results in dysmenorrhea and pelvic pain and often causes infertility. Endometriosis is a significant burden on the quality of life of women. This study will assess the tolerability and how effective elagolix is in changing the disease symptoms in adult female participants with endometriosis.

Elagolix is an approved drug for treatment of endometriosis. Adult female participants with a diagnosis of endometriosis, who are prescribed elagolix by their physicians, in accordance with local clinical practice and label will be observed for up to 24 months. Around 80 female participants will be enrolled in the study in Israel.

Participants will receive Elagolix as prescribed by their physicians.

There may be a higher burden for participants in this study compared to standard of care. Patients report outcomes, in the form of questionnaires will be collected up to 24 months prospectively to assess the impact of elagolix on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with endometriosis and experiencing Dysmenorrhea (DYS).
* Naïve to elagolix prior to starting this study or have stopped taking elagolix for 2 months prior to study enrollment.
* Prescribed elagolix as part of standard treatment for endometriosis, according to the local label.

Exclusion Criteria:

* Contraindication to the use of elagolix.
* Post-menopausal (naturally or surgically).
* Participation in a concurrent interventional clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Female Participants diagnosed with endometriosis and experiencing Dysmenorrhea (DYS).
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Change in Dysmenorrhea (DYS), According to Patient Reported 11-Point Numeric Rating Scale (NRS) | Baseline (Month 0) to Month 3
  Participants rated the change in DYS using an NRS.

SECONDARY OUTCOMES:
Change in Dysmenorrhea (DYS), According to Patient Reported NRS | Baseline (Month 0) through Month 24
  Participants rated the change in DYS using an NRS.
Change in Non-Menstrual Pelvic Pain (NMPP), According to Patient Reported NRS | Baseline (Month 0) through Month 24
  Participants rated the change in NMPP using an NRS.
Change in Dyspareunia, According to Patient Reported NRS | Baseline (Month 0) through Month 24
  Participants rated the change in Dyspareunia using an NRS.
Change in Level of Endometriosis Pain-through Patient Global Impression of Change (PGIC) | Baseline (Month 0) through Month 24
  Participants will evaluate the change in their endometriosis-related pain since initiation of study drug, using the Patient Global Impression of Change (PGIC) questionnaire.
Change in Quality of Life (QoL) through Endometriosis Health Profile-30 (EHP-30) | Baseline (Month 0) through Month 24
  The EHP-30 is a disease-specific self-administered questionnaire used to measure health related QoL in women with endometriosis.
Change in Treatment Satisfaction Though PGIC | Baseline (Month 0) through Month 24
  Participants will evaluate the change in treatment satisfaction through PGIC questionnaire.
Change in Treatment Satisfaction Though Clinician Global Impression of Change (CGIC) | Baseline (Month 0) through Month 24
  The CGIC scale requiring the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
Change in Work Productivity- through Work Productivity and Activity Impairment Questionnaire | Baseline (Month 0) through Month 24
  The Work Productivity and Activity Impairment Questionnaire is used to measure the effect of general health and symptom severity on work productivity and regular activities during the past seven days.
Change in Healthcare Resource Utilization Questionnaire (HCRU) Associated with Endometriosis Through HCRU Questionnaire | Baseline (Month 0) through Month 24
  The HCRU will record the use of health resources (emergency room, physician visit, hospitalization, etc.) prior to and during the study.
Evaluation of Elagolix Dosing | Baseline (Month 0) through Month 24
  Elagolix dosing will be summarized by clinical diagnosis using descriptive statistics including mean, standard deviation, median, quartiles, minimum and maximum and 95% Confidence Interval (CI) for the mean.
Percentage of Participants Who Change Dose of Elagolix | Baseline (Month 0) through Month 24
  Percentage of participants who change dose of elagolix.
Reason Participants Change Dose of Elagolix | Baseline (Month 0) through Month 24
  Reason participants change dose of elagolix.
Percentage of Participants Using Other Treatments of Endometriosis | Baseline (Month 0) through Month 24
  Percentage of participants using other medications or procedures for the treatment of endometriosis.
Percentage of Participants Using Pain/Rescue Medications | Baseline (Month 0) through Month 24
  Percentage of participants using pain/rescue medications.
Percentage of Participants Using Physiotherapy/Cognitive-Behavioral Therapy (Physio/CBT) During and Before the Course of this Observation Period | Baseline (Month 0) through Month 24
  Percentage of participants using physio/CBT during and before the course of this observation period.
Reason for Change at Subsequent Visits in Physiotherapy/Cognitive-Behavioral Therapy (Physio/CBT) During and Before the Course of this Observation Period | Baseline (Month 0) through Month 24
  Reason for change at subsequent visits in physio/CBT during and before the course of this observation period.
Percentage of Participants Using Surgical Intervention During and Before the Course of this Observation Period | Baseline (Month 0) through Month 24
  Percentage of participants using surgical intervention during and before the course of this observation period.
Percentage of Participants Using Add Back | Baseline (Month 0) through Month 24
  Percentage of participants using add back.
Percentage of Participants Using Concomitant Medications | Baseline (Month 0) through Month 24
  Percentage of participants using concomitant medications.
Number of Adverse Events (AEs) | Baseline (Month 0) through Month 24
  An adverse event (AE) is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with their treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- Israel (10):
  - Meir Medical Center /ID# 224766, Kfar Saba, Central District
  - Kaplan Medical Center /ID# 224773, Rehovot, Central District
  - Yitzhak Shamir Medical Center /ID# 224768, Ẕerifin, Central District
  - Hadassah Medical Center-Hebrew University /ID# 224769, Jerusalem, Jerusalem
  - Assuta Ashdod Medical Center /ID# 244898, Ashdod, Southern District
  - Soroka University Medical Center /ID# 224774, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 224764, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 224765, Tel Aviv, Tel Aviv
  - Maccabi Health Services /ID# 224775, Tel Aviv, Tel Aviv
  - Clalit Health Services /ID# 224771, Haifa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related info — https://www.rxabbvie.com
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P20-399#additional-resources-section